CLINICAL TRIAL: NCT00724191
Title: Quantitation of Human Brain Tumor Therapy Response by MR
Brief Title: Evaluation of Human Brain Tumor Therapy Response by Magnetic Resonance (MR)
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas L Chenevert, PhD, Primary Investigator, University of Michigan
Other Study IDs: HUM 00051052; 5P01CA085878-12 (NIH); CA85878-12 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2008-07-24; First posted 2008-07-29 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Evaluation of new MRI methods that measure information related to the chemical makeup of the brain in patients undergoing therapy for brain tumors.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — New MRI methods which measure information related to water, blood, and chemical makeup in the brain.

SUMMARY:
The purpose of this study is to determine if new MRI methods that measure various information and chemical makeup in the brain, will give early information regarding response to treatment in patients with brain tumors.

DETAILED DESCRIPTION:
The purpose of this study is to see if new MRI methods which measure information related to water, blood flow, and chemical makeup in the brain, can give early information of how well treatment is working in patients with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who have been diagnosed with a brain tumor of the central nervous system and a treatment plan has been discussed.
* Must be willing/able to undergo 3-5 MRI scans with IV contrast.
* You can take part in this study if you are NOT afraid of small, enclosed places.

Exclusion Criteria:

* A patient who is claustrophobic.
* Females who are pregnant or lactating.
* Patients who have electrically, magnetically or mechanically activated implants such as heart pacemaker, magnetic surgical clips, prosthesis or or implanted neurological stimulator.
* Any patient who has a history of allergic reactions to MR contrast agent (Omniscan, Magnevist, MultiHance)
* Patients who require general anesthesia to complete MRI exam or patients who have had a negative reaction to MRI sedation. (Chloral Hydrate, Pentobarbital or Versed)
* You should NOT have any metals, or implanted devices in your body (such as aneurysm clips, pacemakers, or artificial joints or limbs.). You will need to tell us about your medical history including any surgeries you have had.

Also, if your job or any other experience might have left metal fragments in your body, please let us know, as the MRI has a strong magnetic field could move a metal fragment in your body or interfere with an implanted device, such as a pacemaker, causing you harm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over of 18 who have been diagnosed with a brain tumor of the central nervous system. Patients must have a treatment plan for their brain tumor from their physician.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 1999-09 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2014-01-15 (Actual)

PRIMARY OUTCOMES:
MRI metrics for brain tumor response | approximately 1 year
  New treatment response MRI metrics derived from change in water diffusion and perfusion from pre-treatment to mid-treatment will be compared to traditional response metrics measured 4 weeks after completion of standard of care chemoradiation for their prediction of patient outcomes and overall survival. The new response metrics are not only measured earlier, but are also quantitative measures for the fraction of tumor exhibiting significant change in diffusion and perfusion assessed on a voxel-by-voxel basis, as well as the volume of dense tumor assessed by analysis of diffusion/perfusion histograms measured over the whole tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Chenevert, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- Univeristy of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No